CLINICAL TRIAL: NCT01968837
Title: The Kilimanjaro Cervical Screening Project
Acronym: KCCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Grand Challenges Canada (Other); Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Principal Investigator, Dr. Karen Yeates, Associate Professor, Department of Medicine, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DMED-1545-12
Record Dates: First submitted 2013-09-30; First posted 2013-10-24 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Uterine Cervical Neoplasms; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cervical cancer screening (No Intervention)
  Interventions: Other: Cervical cancer screening

INTERVENTIONS:
Other: Cervical cancer screening

SUMMARY:
Although highly curable, cervical cancer kills thousands of women in developing countries annually. The investigators will pilot a project to improve detection of cervical cancer in Kilimanjaro, Tanzania through a program that combines access to cervical screening expertise available in a large medical centre and remote use of a mobile phone camera application.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Over 18 years of age

Exclusion Criteria:

* Previous removal of uterus

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1072 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Test accuracy of using digital smart phone cervicograms in place of traditional cervicography images produced through traditional SLR cameras | 3 months

SECONDARY OUTCOMES:
Measure accuracy and feasibility of non-physician healthcare workers ability to obtain adequate cervical images via smart phone camera photographs. | 3 months

OTHER OUTCOMES:
Measure accuracy, quality, and feasibility of SMS text messaging of cervical images obtained by smart phone in place of traditional transfer methods for digital cervical images. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yeates, MD, Principal Investigator — Queen's University
Locations (1):
- Reproductive Health Centre, KCMC, Moshi, Tanzania